CLINICAL TRIAL: NCT02955602
Title: An 8-week, Dose Ranging, Open Label, Randomized, Phase 2 Study With a 44-week Extension, to Evaluate the Safety and Efficacy of MBX-8025 in Subjects With Primary Biliary Cholangitis (PBC) and an Inadequate Response to or Intolerance to Ursodeoxycholic Acid (UDCA)
Brief Title: Seladelpar (MBX-8025) in Subjects With Primary Biliary Cholangitis (PBC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CB8025-21629
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Results first posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-06

CONDITIONS: Primary Biliary Cirrhosis
Keywords: PBC; Primary Biliary Cholangitis (PBC)
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — (2-methyl-4-(5-methyl-2-(4-trifluoromethyl-phenyl)-2H-(1,2,3)triazol-4-ylmethylsulfanyl)phenoxy)acetic acid; seladelpar

ARMS (3):
- MBX-8025 (2 mg) (Experimental): MBX-8025 2 mg capsule once daily
  Interventions: Drug: MBX-8025 2 mg Capsule
- MBX-8025 (5 mg) (Experimental): MBX-8025 5 mg capsule once daily
  Interventions: Drug: MBX-8025 5 mg Capsule
- MBX-8025 (10 mg) (Experimental): MBX-8025 10 mg capsule once daily
  Interventions: Drug: MBX-8025 10 mg Capsule

INTERVENTIONS:
Drug: MBX-8025 2 mg Capsule — Initial 8-week treatment:
  • MBX-8025 2 mg
  Extension:
  The 2 mg group will be started after safety and efficacy review of the 5 mg and the 10 mg groups has been completed.
  Subjects will initially enter the extension on their assigned dose. The dose might be up- or down-titrated after safety and efficacy data review of the first 8 weeks of treatment. During the extension, a subject's dose might be re-adjusted for safety or efficacy reasons.
  Other Names: MBX-8025; seladelpar
  Arms: MBX-8025 (2 mg)
Drug: MBX-8025 5 mg Capsule — Initial 8-week treatment:
  • MBX-8025 5 mg
  Extension:
  Subjects will initially enter the extension on their assigned dose. The dose might be up- or down-titrated after safety and efficacy data review of the first 8 weeks of treatment. During the extension, a subject's dose might be re-adjusted for safety or efficacy reasons.
  Other Names: MBX-8025; seladelpar
  Arms: MBX-8025 (5 mg)
Drug: MBX-8025 10 mg Capsule — Initial 8-week treatment:
  • MBX-8025 10 mg
  Extension:
  Subjects will initially enter the extension on their assigned dose. The dose might be up- or down-titrated after safety and efficacy data review of the first 8 weeks of treatment. During the extension, a subject's dose might be re-adjusted for safety or efficacy reasons.
  Other Names: MBX-8025; seladelpar
  Arms: MBX-8025 (10 mg)

SUMMARY:
An 8-week, dose ranging, open label, randomized, Phase 2 study with a 44-week extension, to evaluate the safety and efficacy of MBX-8025 in subjects with Primary Biliary Cholangitis (PBC) and an inadequate response to or intolerance to ursodeoxycholic acid (UDCA)

DETAILED DESCRIPTION:
Primary:

To evaluate the safety and efficacy of MBX-8025 2 mg, 5 mg, and 10 mg over 8 weeks of treatment

Secondary:

To evaluate the safety and efficacy of MBX-8025 2 mg, 5 mg, and 10 mg over 12 and 26 weeks of treatment

To evaluate the safety and efficacy of MBX-8025 2 mg, 5 mg, and 10 mg over 52 weeks of treatment

To evaluate the pharmacokinetics (PK) of MBX-8025

Exploratory:

To evaluate the effect of MBX-8025 on bile acids, additional markers of inflammation and renal function

MBX-8025 doses of 1 mg and 15 mg may be evaluated if dose adjustment occurs

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent (signed and dated) and any authorizations required by local law
2. 18 to 75 years old (inclusive)
3. Male or female with a diagnosis of PBC, by at least two of the following criteria:

   * History of AP above ULN for at least six months
   * Positive AMA titers (>1/40 on immunofluorescence or M2 positive by enzyme linked immunosorbent assay (ELISA) or positive PBC-specific antinuclear antibodies
   * Documented liver biopsy result consistent with PBC
4. On a stable and recommended dose of UDCA for the past twelve months or intolerant to UDCA
5. AP ≥ 1.67 × ULN
6. Females of reproductive potential must use at least one barrier contraceptive and a second effective birth control method during the study and for at least 90 days after the last dose. Male subjects who are sexually active with female partners of reproductive potential must use barrier contraception and their female partners must use a second effective birth control method during the study and for at least 90 days after the last dose

Exclusion Criteria:

1. A medical condition, other than PBC, that in the investigator's opinion would preclude full participation in the study or confound its results (e.g., cancer on active treatment)
2. AST or ALT > 3 × ULN
3. Total bilirubin > 2.0 mg/dL
4. Total bilirubin > ULN AND albumin < LLN with the exception to subjects with Gilbert's Syndrome. Subjects with Gilbert's syndrome are excluded if Direct Bilirubin > ULN.
5. Auto-immune hepatitis
6. Primary sclerosing cholangitis
7. Known history of alpha-1-Antitrypsin deficiency
8. Known history of chronic viral hepatitis
9. Creatine kinase above ULN
10. Serum creatinine above ULN
11. For females, pregnancy or breast-feeding
12. Use of colchicine, methotrexate, azathioprine, or systemic steroids in the two months preceding screening
13. Current use of fibrates or simvastatin
14. Current use of obeticholic acid
15. Use of an experimental or unapproved treatment for PBC
16. Use of experimental or unapproved immunosuppressant
17. Adverse event leading to MBX-8025 discontinuation from CymaBay's phase 2 PBC study (CB8025-21528)
18. Any other condition(s) that would compromise the safety of the subject or compromise the quality of the clinical study, as judged by the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2019-07-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (23):
  - Institute for Liver Health, Chandler, Arizona
  - Southern California Research Center, Coronado, California
  - Standford University Medicine, Palo Alto, California
  - University of California, Davis Medical Center, Sacramento, California
  - Ventura Clinical Trials, Ventura, California
  - Florida Research Institute, Lakewood Rch, Florida
  - University of Miami - Center for Liver Diseases, Miami, Florida
  - Atlanta Gastroenterology Associates, LLC, Atlanta, Georgia
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Mercy Medical Center, Baltimore, Maryland
  - Henry Ford Health System, Novi, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Louis University, Gastroenterology & Hepatology, St Louis, Missouri
  - Northwell Health - Center for Liver Disease and Transplantation, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - The Mount Sinai Medical Center, New York, New York
  - Northest Clinical Research Center, LLC., Bethlehem, Pennsylvania
  - UT Southwestern Medical Center Investigation Drug Service, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Gastroenterology Consultants of SA, Live Oak, Texas
  - Bon Secours St. Mary's Immaculate Hospital, Newport News, Virginia
  - University of Washington, Seattle, Washington
- Canada (2):
  - University of Calgary Liver Unit, Calgary, Alberta
  - Toronto Centre for Liver Disease, Toronto, Ontario
- Germany (7):
  - Outpatient Clinic of Internal Medicine, Berlin
  - University Hospital Erlangen, Erlangen
  - Ifi-Studien und Projekte GmbH, An der Asklepios Klinik St. Georg, Hamburg
  - Center of Internal Medicine - Medical School of Hannover, Hanover
  - University Medical Centre of the Johannes Guttenberg-University, Mainz
  - Universitatsklinikum Giessen und Marburg GmbH, Marburg
  - Medizinische Universitatsklinik Tubingen, Tübingen
- United Kingdom (6):
  - University Hospitals Birmingham, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Hull and East Yorkshire Hospitals NHS Trust, Hull
  - Royal Free London NHS Foundation Trust, London
  - Plymouth Hospitals NHS Trust, Plymouth
  - Portsmouth Hospitals NHS Trust, Portsmouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bowlus CL, Galambos MR, Aspinall RJ, Hirschfield GM, Jones DEJ, Dorffel Y, Gordon SC, Harrison SA, Kremer AE, Mayo MJ, Thuluvath PJ, Levy C, Swain MG, Neff GW, Sheridan DA, Stanca CM, Berg CP, Goel A, Shiffman ML, Vierling JM, Boudes P, Steinberg A, Choi YJ, McWherter CA. A phase II, randomized, open-label, 52-week study of seladelpar in patients with primary biliary cholangitis. J Hepatol. 2022 Aug;77(2):353-364. doi: 10.1016/j.jhep.2022.02.033. Epub 2022 Mar 30. PMID 35367282

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 192 subjects were screened of which 121 subjects randomized (2 subjects were not treated) into the study and 71 were screen failures. Subjects were randomized to the 5 and 10 mg treatment groups for entry to the 8-week initial treatment period study, while those in the 2 mg treatment group entered after being sequentially assigned their dose
Groups:
- MBX-8025 (2 mg): MBX-8025 2 mg capsule once daily
  MBX-8025 2 mg Capsule: Initial 8-week treatment:
  • MBX-8025 2 mg
  Subjects received two seladelpar 1 milligram (mg) capsules orally once daily for 8 weeks with a 44-week extension period. Dose up-titration for efficacy reasons could be made after 12 weeks of treatment up to 10 mg.
- MBX-8025 (5 mg): MBX-8025 5 mg capsule once daily
  MBX-8025 5 mg Capsule: Initial 8-week treatment:
  • MBX-8025 5 mg
  Subjects were randomized to receive one seladelpar 5 mg capsule orally once daily for 8 weeks with a 44-week extension period. Dose up-titration to 10 mg for efficacy reasons could be made after 12 weeks of treatment.
- MBX-8025 (10 mg): MBX-8025 10 mg capsule once daily
  MBX-8025 10 mg Capsule: Initial 8-week treatment:
  • MBX-8025 10 mg
  Subjects were randomized to receive one seladelpar 10 mg capsule orally once daily for 8 weeks with a 44-week extension period.
Period: Overall Study
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Started | 11 | 53 | 55
Completed | 10 | 46 | 49
Not Completed | 1 | 7 | 6
Not completed — Adverse Event | 0 | 3 | 0
Not completed — Withdrawal of informed consent | 1 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Other | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: 18 to 75 years of age (inclusive)
Groups:
- Total: Total of all reporting groups
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg) | Total
Number analyzed (Participants) | 11 | 53 | 55 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 41 | 41 | 90
  >=65 years | 3 | 12 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (9.6) | 57.5 (8.1) | 57.4 (9.7) | 56.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 51 | 50 | 112
  Male | 0 | 2 | 5 | 7
Race/Ethnicity, Customized [Number; unit: Subjects]
  White | 10 | 50 | 49 | 109
  Black or African-American | 0 | 1 | 3 | 4
  Asian | 0 | 2 | 1 | 3
  American Indian or Alaska native | 0 | 0 | 1 | 1
  Other | 1 | 0 | 0 | 1
  Multiple | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 5 | 1 | 6
  United States | 0 | 39 | 43 | 82
  United Kingdom | 11 | 5 | 4 | 20
  Germany | 0 | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Relative Change From Baseline in Serum Alkaline Phosphatase (ALP) at Week 8
Description: Relative change from baseline in serum ALP levels at Week 8 (endpoint). The modified Intent-to-Treat (mITT) analysis set included all randomized subjects with confirmed PBC who received at least one study drug dose and had at least one post baseline ALP evaluation on treatment. n, denotes number of subjects evaluable for the respective timepoints
Time Frame: 8 weeks
Population: mITT Population The mITT population is defined as any enrolled subject who receives at least one dose of medication and has at least one post-baseline AP evaluation and who have confirmed PBC.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 47 | 51
percentage change from baseline | -26.06 (9.15) | -33.38 (17.81) | -41.42 (13.05)
Statistical Analysis 1: Comparison: MBX-8025 (2 mg) vs MBX-8025 (5 mg); The analyses will assess the change from baseline in each treatment group and will assess the hypothesis that there are no differences in the percent change in ALP serum level between seladelpar 2 mg and 5 mg treatment groups after 8 weeks of treatment; Test type: Other; p = 0.2242, ANCOVA
Statistical Analysis 2: Comparison: MBX-8025 (2 mg) vs MBX-8025 (10 mg); The analyses will assess the change from baseline in each treatment group and will assess the hypothesis that there are no differences in the percent change in ALP serum level between seladelpar 2 mg and 10 mg treatment groups after 8 weeks of treatment; Test type: Other; p = 0.0021, ANCOVA
Statistical Analysis 3: Comparison: MBX-8025 (5 mg) vs MBX-8025 (10 mg); The analyses will assess the change from baseline in each treatment group and will assess the hypothesis that there are no differences in the percent change in ALP serum level between seladelpar 5 mg and 10 mg treatment groups after 8 weeks of treatment; Test type: Other; p = 0.0024, ANCOVA

2. Secondary Outcome: Absolute Change From Baseline in Serum Alkaline Phosphatase (ALP) at Week 12 and Week 52
Description: Absolute change in ALP from baseline to Weeks 12 and 52 The mITT analysis set included all randomized subjects with confirmed PBC who received at least one study drug dose and had at least one post baseline ALP evaluation on treatment.
Time Frame: 12 weeks and 52 weeks
Population: mITT Population: The mITT population is defined as any enrolled subject who receives at least one dose of medication and has at least one post-baseline AP evaluation and who have confirmed PBC.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 49 | 52
U/L
  Absolute Change at Week 12: number analyzed (Participants) | 11 | 46 | 49
  Absolute Change at Week 12 | -68.318 (63.276) | -135.902 (150.954) | -127.867 (60.284)
  Absolute Change at Week 52: number analyzed (Participants) | 10 | 42 | 48
  Absolute Change at Week 52 | -101.150 (107.956) | -158.310 (143.668) | -133.760 (76.151)

3. Secondary Outcome: Change in Aspartate Aminotransferase (AST) From Baseline to 12 Weeks and 52 Weeks
Description: Change from baseline in AST levels at endpoint was reported. The mITT analysis set included all randomized subjects with confirmed PBC who received at least one study drug dose and had at least one post baseline ALP evaluation on treatment.
Time Frame: 12 weeks and 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 49 | 52
U/L
  Week 12: number analyzed (Participants) | 11 | 46 | 49
  Week 12 | -2.50 (16.72) | -1.13 (24.28) | -3.35 (10.55)
  Week 52: number analyzed (Participants) | 10 | 42 | 48
  Week 52 | -7.05 (10.50) | -6.18 (13.98) | -6.14 (9.18)

4. Secondary Outcome: Change in Alanine Aminotransferase (ALT) From Baseline to 12 Weeks and 52 Weeks
Description: Change from baseline in ALT levels at endpoint was reported. The mITT analysis set included all randomized subjects with confirmed PBC who received at least one study drug dose and had at least one post baseline ALP evaluation on treatment.
Time Frame: 12 weeks and 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 49 | 52
U/L
  Week 12: number analyzed (Participants) | 11 | 46 | 49
  Week 12 | -5.59 (16.07) | -10.48 (21.41) | -10.87 (20.25)
  Week 52: number analyzed (Participants) | 10 | 42 | 48
  Week 52 | -14.30 (25.12) | -17.29 (17.46) | -15.32 (13.89)

5. Secondary Outcome: Change in Gamma-glutamyl Transferase (GGT) From Baseline to 12 Weeks and 52 Weeks
Description: Change from baseline in GGT levels at endpoint was reported. The mITT analysis set included all randomized subjects with confirmed PBC who received at least one study drug dose and had at least one post baseline ALP evaluation on treatment.
Time Frame: 12 weeks and 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 49 | 52
U/L
  Week 12: number analyzed (Participants) | 11 | 46 | 49
  Week 12 | -43.68 (56.87) | -75.35 (87.57) | -80.82 (109.06)
  Week 52: number analyzed (Participants) | 10 | 42 | 48
  Week 52 | -78.60 (81.59) | -91.37 (102.23) | -88.08 (122.14)

6. Secondary Outcome: Change in Bilirubin - Total Bilirubin (TB) From Baseline to 12 Weeks and 52 Weeks
Description: Change from baseline in TB levels at endpoint is being reported. The mITT analysis set included all randomized subjects with confirmed PBC who received at least one study drug dose and had at least one post baseline ALP evaluation on treatment.
Time Frame: 12 weeks and 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 49 | 52
mg/dL
  Week 12: number analyzed (Participants) | 11 | 46 | 49
  Week 12 | -0.010 (0.121) | -0.055 (0.161) | -0.067 (0.199)
  Week 52: number analyzed (Participants) | 10 | 42 | 48
  Week 52 | 0.002 (0.152) | -0.028 (0.263) | -0.068 (0.190)

7. Secondary Outcome: Percentage of Participants Meet Composite Endpoint Criteria of ALP and Total Bilirubin
Description: Participant meets composite endpoint is defined by participant meets all of the following criteria:
  * ALP < 1.67 × upper limit of normal (ULN)
  * Total Bilirubin within normal limit
  * > 15% decrease in ALP
  Endpoint of Alkaline Phosphatase and Total Bilirubin by Visit (mITT Population)
Time Frame: 12 Weeks and 52 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 49 | 52
percentage of participants
  Week 12: number analyzed (Participants) | 11 | 47 | 51
  Week 12 | 45.5 | 48.9 | 66.7
  Week 52: number analyzed (Participants) | 11 | 45 | 49
  Week 52 | 63.6 | 53.3 | 67.3

8. Secondary Outcome: Percentage of Participants Meet Published PBC Response Criteria - Paris I
Description: Percentage of participants with response based on Paris I risk score was defined as ALP less than or equal to (≤) 3x ULN and aspartate aminotransferase (AST) less than or equal to (≤) 2 x ULN and Total Bilirubin ≤ 1 mg/dL.
  The mITT analysis set included all randomized subjects with confirmed PBC who received at least one study drug dose and had at least one post baseline ALP evaluation on treatment.
Time Frame: 12 weeks and 52 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 49 | 52
percentage of participants
  Week 12: number analyzed (Participants) | 11 | 46 | 49
  Week 12 | 81.8 | 76.1 | 75.5
  Week 52: number analyzed (Participants) | 10 | 42 | 48
  Week 52 | 90 | 81.0 | 79.2

9. Secondary Outcome: Percentage of Participants Meet Published PBC Response Criteria - Paris II
Description: Percentage of participants with response based on Paris II risk score was defined as ALP≤1.5xULN and AST≤1.5xULN and Total Bilirubin ≤ 1 mg/dL.
  The mITT analysis set included all randomized subjects with confirmed PBC who received at least one study drug dose and had at least one post baseline ALP evaluation on treatment.
Time Frame: 12 weeks and 52 weeks
Population: mITT Population. The mITT population is defined as any enrolled subject who receives at least one dose of medication and has at least one post-baseline AP evaluation and who have confirmed PBC.
Measure: Number; unit: percentage of participants
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 49 | 52
percentage of participants
  Week 12: number analyzed (Participants) | 11 | 46 | 49
  Week 12 | 36.4 | 37.0 | 59.2
  Week 52: number analyzed (Participants) | 10 | 42 | 48
  Week 52 | 50.0 | 54.8 | 60.4

10. Secondary Outcome: Percentage of Participants Meet Published PBC Response Criteria - Toronto I
Description: Percentage of participants with response based on Toronto I risk score defined as ALP ≤ 1.67 x ULN. The mITT analysis set included all randomized subjects with confirmed PBC who received at least one study drug dose and had at least one post baseline ALP evaluation on treatment.
Time Frame: 12 weeks and 52 weeks
Population: as for outcome 9
Measure: Number; unit: percentage of subjects
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 49 | 52
percentage of subjects
  Week 12: number analyzed (Participants) | 11 | 47 | 51
  Week 12 | 63.6 | 51.1 | 78.4
  Week 52: number analyzed (Participants) | 11 | 45 | 49
  Week 52 | 63.6 | 57.8 | 71.4

11. Secondary Outcome: UK-PBC Risk Score Value
Description: The UK-PBC Risk Score at endpoint is defined by the mean percentage risk that a PBC patient treated with ursodeoxycholic acid (UDCA) would develop liver failure requiring liver transplantation in 5, 10 and 15 years from diagnosis. The higher the score might indicate higher risk to death or live transplantation. Formula used for UK-PBC risk score = 1- 0.982 ^EXP(0.0287854*(ALP12 x ULN-1.722136304) - 0.0422873*(((TA12 xULN/10)^-1) - 8.675729006) + 1.4199 * (LN(BIL12 x ULN/10)+2.709607778)-1.960303*(Albumin x LLN-1.17673001)-0.4161954*(Platelet x LLN-1.873564875)). Where, Baseline survivor function = 0.982, 0.941, and 0.893 for 5 years, 10 years and 15 years respectively. ALP12, TA12 and BIL12 refers to the ALP, transaminases (ALT, AST), and total bilirubin assessments, respectively. The modified Intent-to-Treat (mITT) analysis set included all randomized subjects with confirmed PBC who received at least one study drug dose and had at least one post baseline ALP evaluation on treatment.
Time Frame: 12 weeks and 52 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 49 | 52
units on a scale
  5 years, week 12: number analyzed (Participants) | 11 | 44 | 48
  5 years, week 12 | 1.3929 (0.6976) | 2.2553 (2.5145) | 1.8124 (1.7267)
  5 years, week 52: number analyzed (Participants) | 10 | 40 | 47
  5 years, week 52 | 1.3145 (0.7704) | 2.3485 (3.432) | 1.7244 (1.6121)
  10 years week 12: number analyzed (Participants) | 11 | 44 | 48
  10 years week 12 | 4.5705 (2.2479) | 7.1229 (7.4904) | 5.8293 (5.3605)
  10 years, week 52: number analyzed (Participants) | 10 | 40 | 47
  10 years, week 52 | 4.3128 (2.4649) | 7.2322 (9.5794) | 5.5607 (5.0092)
  15 years, week 12: number analyzed (Participants) | 11 | 44 | 48
  15 years, week 12 | 8.3008 (3.9932) | 12.4002 (12.1785) | 10.3469 (9.1269)
  15 years, week 52: number analyzed (Participants) | 10 | 40 | 47
  15 years, week 52 | 7.8325 (4.3413) | 12.3028 (14.5701) | 9.9008 (8.5396)

12. Secondary Outcome: Change From Baseline in Pruritus Visual Analog Score (VAS) at Week 12 and Week 52
Description: VAS is the commonly used graphic tool for self-reporting of pruritus intensity in patients. VAS is a simple to use, validated, reliable and widely applicable tool that does not determine the impact of pruritus to quality of life. It comprises of a 100-mm horizontal line labelled as "no symptom" on left end and "worst imaginable symptom" on right end. Based on the intensity of the itch patient is instructed to draw a vertical line on the horizontal scale having a range [VAS values (unit: mm) ranging from 0 to 100, where 0 represents "no itching" and 100 "worst possible itching"].
  The modified Intent-to-Treat (mITT) analysis set included all randomized subjects with confirmed PBC who received at least one study drug dose and had at least one post baseline ALP evaluation on treatment.
Time Frame: 12 weeks and 52 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 49 | 52
score on a scale
  Week 12: number analyzed (Participants) | 11 | 45 | 49
  Week 12 | -3.7 (6.4) | -5.5 (25.0) | -12.3 (22.3)
  Week 52: number analyzed (Participants) | 10 | 42 | 48
  Week 52 | -3.3 (11.7) | -9.6 (22.5) | -16.5 (23.0)

13. Secondary Outcome: Change From Baseline in PBC-40 Quality of Life (QoL) at Week 12 and Week 52
Description: The PBC-40 QoL questionnaire is a disease-specific health-related tool developed for measuring the psychometric profile in PBC patients. It has 10 domains and 43 questions relevant to PBC, including Cognitive, Social, Emotional Function, Fatigue, Itch, and Other Symptoms. Questions in domains: 1) digestion and diet (questions 1-3); 2) experiences (questions 4-7); 3) itching (questions 8-10); 4) fatigue (questions 11-18); 5) effort and planning (questions 19-21); 6) memory and concentration (questions 22-27); 7) affects to you as person (questions 28-33); 8) affects to your social life (questions 34-37); 9) overall impact on your life (questions 38-40); 10) general health and well-being (questions A-C). Within a domain, items are scored from 1 to 5 and the individual item scores are summed to give a total domain score. High scores represent high impact and low scores low impact of PBC on QoL (mITT Population).
Time Frame: 12 weeks and 52 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 49 | 52
units on a scale
  General Symptoms, Week 12: number analyzed (Participants) | 11 | 45 | 49
  General Symptoms, Week 12 | 1.9 (2.7) | -0.7 (5.1) | -0.5 (3.6)
  General Symptoms, Week 52: number analyzed (Participants) | 10 | 42 | 48
  General Symptoms, Week 52 | 0.3 (2.4) | -1.4 (4.4) | -0.1 (4.4)
  Itch, Week 12: number analyzed (Participants) | 11 | 45 | 49
  Itch, Week 12 | -0.4 (2.0) | -0.5 (3.4) | -0.8 (3.1)
  Itch, Week 52: number analyzed (Participants) | 10 | 42 | 48
  Itch, Week 52 | 0.4 (2.7) | -1.3 (3.2) | -1.4 (3.7)
  Fatigue, Week 12: number analyzed (Participants) | 11 | 45 | 49
  Fatigue, Week 12 | -1.5 (6.1) | -2.1 (10.4) | -3.0 (5.2)
  Fatigue, Week 52: number analyzed (Participants) | 10 | 42 | 48
  Fatigue, Week 52 | -1.2 (7.8) | -3.0 (8.5) | -3.4 (6.3)
  Cognitive Function, Week 12: number analyzed (Participants) | 11 | 45 | 49
  Cognitive Function, Week 12 | -0.9 (2.4) | -0.6 (5.7) | -0.7 (2.8)
  Cognitive Function, Week 52: number analyzed (Participants) | 10 | 42 | 48
  Cognitive Function, Week 52 | -0.7 (7.6) | -1.4 (5.3) | -0.6 (2.5)
  Social, Week 12: number analyzed (Participants) | 11 | 44 | 49
  Social, Week 12 | 0.8 (2.8) | -0.5 (7.9) | -1.0 (6.3)
  Social, Week 52: number analyzed (Participants) | 10 | 42 | 48
  Social, Week 52 | -3.3 (5.2) | -1.6 (7.2) | -1.6 (6.2)
  Emotional, Week 12: number analyzed (Participants) | 11 | 44 | 48
  Emotional, Week 12 | -0.9 (1.6) | -1.0 (2.6) | -0.8 (2.1)
  Emotional, Week 52: number analyzed (Participants) | 10 | 42 | 47
  Emotional, Week 52 | -2.1 (2.3) | -1.3 (2.7) | -0.9 (2.1)

14. Secondary Outcome: Percentage of Participants Meet Published PBC Response Criteria - Barcelona
Description: Percentage of participants with response based on Barcelona risk scores was defined as Normalization of ALP or a Decrease of ALP ≥ 40%. The mITT analysis set included all randomized subjects with confirmed PBC who received at least one study drug dose and had at least one post baseline ALP evaluation on treatment.
Time Frame: 12 weeks and 52 weeks
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 49 | 52
percentage of participants
  Week 12: number analyzed (Participants) | 11 | 47 | 51
  Week 12 | 9.1 | 42.6 | 62.7
  Week 52: number analyzed (Participants) | 11 | 45 | 49
  Week 52 | 45.5 | 66.7 | 65.3

15. Secondary Outcome: Absolute Change in MELD Score From Baseline to 12 Weeks and 52 Weeks
Description: Change from baseline to 12 weeks and 52 weeks in Model for End-stage Liver Disease (MELD) Score (mITT Population) The MELD score ranges from 6 to 40 and is a measure of how severe a patient's liver disease is. The higher the score, the more likely the patients will need a liver transplant. A calculated prognostic risk factor used to assess the potential need for a liver transplant.
  MELD(i) score = 10*[0.957*ln(creatinine mg/dL) + 0. 378*ln(total bilirubin mg/dL) + 1.120*ln (INR) + 0.643].
  If MELD(i) is less than or equal to 11 then MELD = MELD(i). If MELD(i) is greater than 11 then MELD = MELD(i) + (1.32 *(137 - (Na)) - (0.033*MELD(i)*(137 - Na))
Time Frame: 12 weeks and 52 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Change from Baseline
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 49 | 52
Change from Baseline
  Week 12: number analyzed (Participants) | 11 | 46 | 48
  Week 12 | -0.3 (1.6) | 0.1 (1.2) | 0.1 (1.0)
  Week 52: number analyzed (Participants) | 10 | 42 | 48
  Week 52 | -0.7 (1.6) | 0.3 (1.1) | 0.2 (1.2)

16. Secondary Outcome: Change in GLOBE PBC Score From Baseline to 12 Weeks and 52 Weeks
Description: Change from Baseline to 12 weeks and 52 weeks in Global PBC Study Group (GLOBE) score (mITT Population)
  The GLOBE score is a validated risk assessment tool providing an estimate of transplant-free survival for patients with PBC. It was developed by the Global PBC Study Group using Cox regression model on over 4,000 patients with PBC. Lower GLOBE score predicts lower risk. It is calculated from the following equation:
  GLOBE score = (0.044378 * age + 0.93982 * LN(total bilirubin/ULN) +(0.335648 * LN(alkaline phosphatase/ULN)) - 2.266708 * albumin /LLN -0.002581 * platelet count per 109/L) + 1.216865
Time Frame: 12 weeks and 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 49 | 52
units on a scale
  Week 12: number analyzed (Participants) | 10 | 43 | 46
  Week 12 | -0.079 (0.260) | -0.292 (0.304) | -0.346 (0.269)
  Week 52: number analyzed (Participants) | 9 | 37 | 43
  Week 52 | -0.180 (0.217) | -0.271 (0.354) | -0.404 (0.298)

17. Secondary Outcome: Participants Meet Rotterdam Criteria
Description: participants with Response Based on Rotterdam Criteria at Weeks 12 and 52 Rotterdam Published PBC Response Criteria by Visit (mITT Population) Rotterdam criteria: Early (normal total bilirubin and normal albumin), Moderately advanced (either abnormal albumin or abnormal total bilirubin), and Advanced (both abnormal albumin and abnormal total bilirubin). From Early stage to Moderate Stage and to Advanced Stage, it becomes worse and worse in abnormality.
Time Frame: 12 weeks and 52 weeks
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 49 | 52
participants
  Early Stage,12 Weeks: number analyzed (Participants) | 11 | 46 | 49
  Early Stage,12 Weeks | 11 | 38 | 40
  Early Stage, 52 weeks: number analyzed (Participants) | 10 | 42 | 48
  Early Stage, 52 weeks | 10 | 36 | 42
  Moderately advanced at 12 Weeks: Either abnormal Albumin or abnormal Total Bilirubin: number analyzed (Participants) | 11 | 46 | 49
  Moderately advanced at 12 Weeks: Either abnormal Albumin or abnormal Total Bilirubin | 0 | 7 | 9
  Moderately advanced: 52 Weeks, Either abnormal Albumin or abnormal Total Bilirubin: number analyzed (Participants) | 10 | 42 | 48
  Moderately advanced: 52 Weeks, Either abnormal Albumin or abnormal Total Bilirubin | 0 | 3 | 5
  Advanced: 12 Weeks, Both abnormal Albumin and abnormal Total Bilirubin: number analyzed (Participants) | 11 | 46 | 49
  Advanced: 12 Weeks, Both abnormal Albumin and abnormal Total Bilirubin | 0 | 1 | 0
  Advanced: 52 Weeks Both abnormal Albumin and abnormal Total Bilirubin: number analyzed (Participants) | 10 | 42 | 48
  Advanced: 52 Weeks Both abnormal Albumin and abnormal Total Bilirubin | 0 | 3 | 1

18. Secondary Outcome: Percentage of Participants Meet Composite Endpoint of AP and Total Bilirubin Criteria at Week 12 and Week 52
Description: Percentage of participants with Response Defined by Composite Endpoint (ALP< 1.67 * Upper Limit of Normal [ULN] at Endpoint, Total Bilirubin [BIL] within Normal Limits at Endpoint, and Greater Than Equal To [≥] 15% ALP Reduction) from Baseline to Week 12 and Week 52 The mITT analysis set included all randomized subjects with confirmed PBC who received at least one study drug dose and had at least one post baseline ALP evaluation on treatment.
Time Frame: 12 weeks and 52 weeks
Population: as for outcome 9
Measure: Number; unit: percentage of subjects
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 49 | 52
percentage of subjects
  Week 12: number analyzed (Participants) | 11 | 47 | 51
  Week 12 | 45.5 | 48.9 | 66.7
  Week 52: number analyzed (Participants) | 11 | 45 | 49
  Week 52 | 63.6 | 53.3 | 67.3

19. Secondary Outcome: Percent Change in Serum Alkaline Phosphatase (ALP)
Description: Percent change in ALP from baseline to Weeks 12 and 52 The mITT analysis set included all randomized subjects with confirmed PBC who received at least one study drug dose and had at least one post baseline ALP evaluation on treatment.
Time Frame: 12 weeks and 52 weeks
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage Change
Arm/Group | MBX-8025 (2 mg) | MBX-8025 (5 mg) | MBX-8025 (10 mg)
Number analyzed (Participants) | 11 | 49 | 52
percentage Change
  Relative Change at Week 12: number analyzed (Participants) | 11 | 47 | 51
  Relative Change at Week 12 | -22.56 (13.92) | -34.49 (20.62) | -43.20 (12.39)
  Relative Change at Week 52: number analyzed (Participants) | 11 | 45 | 49
  Relative Change at Week 52 | -32.72 (22.48) | -40.09 (24.23) | -44.19 (15.52)

ADVERSE EVENTS:
Time Frame: Up to Week 56
Groups:
- MBX-8025 2 mg: MBX-8025 2 mg capsule once dailyMBX-8025 2 mg Capsule: Initial 8-week treatment:• MBX-8025 2 mgSubjects received two seladelpar 1 milligram (mg) capsules orally once daily for 8 weeks with a 44-week extension period. Dose up-titration for efficacy reasons could be made after 12 weeks of treatment up to 10 mg
- MBX-8025 5 mg: MBX-8025 5 mg capsule once dailyMBX-8025 5 mg Capsule: Initial 8-week treatment:• MBX-8025 5 mgSubjects were randomized to receive one seladelpar 5 mg capsule orally once daily for 8 weeks with a 44-week extension period. Dose up-titration to 10 mg for efficacy reasons could be made after 12 weeks of treatment.
- MBX-8025 10 mg: MBX-8025 10 mg capsule once dailyMBX-8025 10 mg Capsule: Initial 8-week treatment:• MBX-8025 10 mgSubjects were randomized to receive one seladelpar 10 mg capsule orally once daily for 8 weeks with a 44-week extension period.
Arm/Group | MBX-8025 2 mg | MBX-8025 5 mg | MBX-8025 10 mg
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/53 | 0/55
Serious Adverse Events (participants affected / at risk) | 1/11 | 8/53 | 5/55
Other Adverse Events (participants affected / at risk) | 11/11 | 45/53 | 47/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MBX-8025 2 mg (N=11) | MBX-8025 5 mg (N=53) | MBX-8025 10 mg (N=55)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pyonephrosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MBX-8025 2 mg (N=11) | MBX-8025 5 mg (N=53) | MBX-8025 10 mg (N=55)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2)
Dry eye (Eye disorders) | 2 (2) | 1 (1) | 4 (4)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 4 (4) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 7 (8) | 5 (5)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 7 (7) | 9 (9)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4)
Dyschezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (4) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 5 (7) | 5 (5)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (8) | 9 (11) | 6 (6)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (6) | 5 (5)
Asthenia (General disorders) | 1 (2) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (2) | 0 (0)
Fatigue (General disorders) | 3 (3) | 9 (10) | 6 (6)
Feeling of body temperature change (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (3) | 2 (2)
Peripheral swelling (General disorders) | 1 (1) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 2 (2)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Allergy to vaccine (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3) | 3 (3)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 5 (5) | 2 (2)
Nasopharyngitis (Infections and infestations) | 4 (5) | 5 (7) | 6 (9)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 5 (6) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (2) | 8 (11) | 8 (12)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 4 (4)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (6) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 5 (5) | 3 (3)
Headache (Nervous system disorders) | 2 (5) | 6 (9) | 3 (3)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (5) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (9) | 11 (13) | 12 (12)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
First, there was an imbalance in baseline ALP levels among cohorts. Second, the criteria for dose uptitration were not standardized, except that uptitration could only be done at or after Week 12. Third, this was not a placebo-controlled study. Finally, multiplicity adjustments were not made for efficacy endpoints. Nominal p-values were provided for descriptive purposes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT02955602/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT02955602/SAP_001.pdf